CLINICAL TRIAL: NCT00159653
Title: A 12-Week, Randomized, Double-Masked, Parallel Group Comparison Of Xalacom Given In The Evening, Xalatan Given In The Evening, And Timolol Given In The Morning In Patients With Open Angle Glaucoma Or Ocular Hypertension.
Brief Title: A 12-Week, Randomized, Double-Masked, Parallel Group Comparison Of Evening Dosing With Xalacom In Subjects With Glaucoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6641027
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2012-10

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Xalacom; Latanoprost; Timolol

INTERVENTIONS:
Drug: Xalacom
Drug: Xalatan
Drug: Timolol

SUMMARY:
To demonstrate statistical superiority of the combination of latanoprost and timolol to the individual therapy of latanoprost and timolol based on intraocular pressure measurements at 8 AM, 10 AM, 4 PM at weeks 2, 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Uni- or bilateral diagnosis of primary open angle glaucoma or ocular hypertension on beta-blocker monotherapy or dual therapy in which at least one medication is a beta-blocker for at least 4 weeks prior to screening

Exclusion Criteria:

* Closed/ barely open anterior chamber angle or history of acute angle closure glaucoma.
* History of ALT (Argon Laser Trabeculoplasty) or SLT(selective Laser) within 3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2005-07; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The mean IOP measurements obtained in the study eye at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- United States (33):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Poway, California
  - Pfizer Investigational Site, Redding, California
  - Pfizer Investigational Site, Danbury, Connecticut
  - Pfizer Investigational Site, Cape Coral, Florida
  - Pfizer Investigational Site, Lakeland, Florida
  - Pfizer Investigational Site, Ormond Beach, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Morrow, Georgia
  - Pfizer Investigational Site, Homewood, Illinois
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, North Dartmouth, Massachusetts
  - Pfizer Investigational Site, Saint Joseph, Michigan
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Newark, New Jersey
  - Pfizer Investigational Site, Bethpage, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, High Point, North Carolina
  - Pfizer Investigational Site, Matthews, North Carolina
  - Pfizer Investigational Site, Wilmington, North Carolina
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Cranberry Township, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, North Charleston, South Carolina
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Amarillo, Texas
  - Pfizer Investigational Site, Houston, Texas
- Canada (12):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Nanaimo, British Columbia
  - Pfizer Investigational Site, Moncton, New Brunswick
  - Pfizer Investigational Site, Saint John, New Brunswick
  - Pfizer Investigational Site, Bridgewater, Nova Scotia
  - Pfizer Investigational Site, Barrie, Ontario
  - Pfizer Investigational Site, Markham, Ontario
  - Pfizer Investigational Site, Mississauga, Ontario
  - Pfizer Investigational Site, Oakville, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Saskatoon, Saskatchewan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6641027&StudyName=A%2012-Week%2C%20Randomized%2C%20Double-Masked%2C%20Parallel%20Group%20Comparison%20Of%20Evening%20Dosing%20With%20Xalacom%20In%20Subjects%20With%20Glaucoma